CLINICAL TRIAL: NCT06165198
Title: Individualized Neuromodulation Intervention Techniques for the Core Clinical Features of Drug Addiction
Brief Title: Individualized Neuromodulation for the Core Clinical Features of Drug Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZhao-013
Record Dates: First submitted 2023-09-16; First posted 2023-12-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2023-09

CONDITIONS: Amphetamine Use Disorders
Keywords: individualized therapy; closed-loop; Amphetamine-type stimulants; tACS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop tACS stimulation based on addiction-induced states (Experimental): In the initial phase of this study, participants will be subjected to individual closed-loop tACS interventions at varying frequencies for one-week intervals. Concurrently, they will be exposed to MA-related cue paradigms to induce brain addiction states, while scalp EEG signals are collected. Stimulation will be initiated only upon identifying specific neural signals associated with MA cues, aiming to ascertain the optimal frequency for single-session closed-loop tACS stimulation that could elicit individual neurological responses. Subsequently, we will embark on a longitudinal closed-loop tACS intervention control study for MA dependents at one-week intervals, which involves addiction-induced closed-loop tACS stimulation, random time-point stimulation, and traditional continuous stimulation, to rectify potential sequence effects and delineate the disparities in neurological and behavioral impacts between discrete and continuous stimulations based on brain states.
  Interventions: Device: Closed-loop tACS stimulation based on addiction-induced states

INTERVENTIONS:
Device: Closed-loop tACS stimulation based on addiction-induced states — We conducted a longitudinal controlled study of closed-loop tACS interventions among MA dependents.This involved implementing interventions based on addiction-induced states through closed-loop tACS stimulation, randomized time-point stimulation, and traditional continuous stimulation.

SUMMARY:
Using specific EEG biomarkers in methamphetamine-dependent individuals, this study systematically probes closed-loop tACS based on brain states, assessing dosage, neurologic and behavioral effects, while comparing its efficacy with traditional open-loop tACS methods.

DETAILED DESCRIPTION:
The current study delineates a robust correlation between prefrontal cortex EEG signals and the psychological craving associated with methamphetamine usage. Dependents exhibit heightened β oscillation energy in the MPFC region and diminished γ oscillation energy across the DLPFC-MPFC region. Previously, through the implementation of rTMS interventions on the left DLPFC, the investigators have successfully reduced the craving levels in users when exposed to relevant cues, coupled with observed decreases in β oscillation energy and increases in γ oscillation energy in the MPFC region. This indicates that both β and γ oscillation energies are instrumental in representing the involvement of MPFC and DLPFC during craving episodes, and neuromodulatory technologies can modulate these energy levels, consequently reducing cravings. Furthermore, the investigators identified a significant augmentation in the theta energy in the occipital lobe when MA dependents are confronted with drug-related cue imagery, signifying a potential crucial neural marker for addiction-induced brain activity. Therefore, the investigators intend to employ the non-invasive transcranial alternating current stimulation (tACS) technique, predicated upon biomarkers of addiction states, to administer specific frequency stimulations to targeted brain regions, aiming to achieve therapeutic objectives in addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 45 years, irrespective of gender, having completed a minimum of 9 years of education and capable of effectively cooperating in questionnaire evaluations.
* Meet the diagnostic criteria set forth by the DSM-V concerning the severity of amphetamine-type substance addiction.
* A history of utilizing amphetamine-type substances for a duration not less than one year, with a frequency of use being at least once per week.
* Consent to actively cooperate in the completion of subsequent follow-up assessments.

Exclusion Criteria:

* Severe cognitive functional impairments manifested through a history of head trauma, cerebrovascular diseases, epilepsy, etc., or usage of cognitive enhancement drugs in the past 6 months; an intellectual disability with an IQ score less than 70.
* A diagnosis of schizophrenia or other severe mental illnesses as per the DSM-5 criteria.
* Abuse or dependence on other psychoactive substances (excluding nicotine) within the past 5 years.
* Severe organic diseases that might compromise study participation.
* Contraindications to tACS, such as a history of epileptic seizures or the presence of metallic implants in proximity to the head.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Stop-signal task | through study completion, an average of 1 month
  The stop-signal task can indicate executive control capabilities by measuring Stop-signal reaction time, Stop-signal delays, Go-task reaction time, and Success and failure inhibition rates.

SECONDARY OUTCOMES:
Changes of electroencephalogram power spectrum | through study completion, an average of 1 month
  Resting-state EEG can be used to extract power spectra and electrode functional connectivity; on-task EEG can be used to isolate time-frequency features during non-stimulated trials to extract alpha, beta, theta, and gamma band energy of the parietal and occipital electrodes. Both can be used to assess changes in neural activity before, during, and after their restimulation.

CONTACTS AND LOCATIONS:
Overall Officials: MIn Zhao, PhD, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No